CLINICAL TRIAL: NCT01869803
Title: Compassionate Use of Gemtuzumab Ozogamicin (Mylotarg) for Treatment of Patients With Relapsed or Refractory CD33-Positive Acute Myeloid Leukemia (AML) or Acute Promyelocytic Leukemia (APL)
Brief Title: Gemtuzumab Ozogamicin in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia or Acute Promyelocytic Leukemia
Status: Approved for marketing | Type: Expanded Access
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CCCWFU# 99213; NCI-2013-00965 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA012197 (NIH)
Record Dates: First submitted 2013-05-31; First posted 2013-06-05 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Promyelocytic Leukemia (M3); Childhood Acute Promyelocytic Leukemia (M3); Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Promyelocytic, Acute; Leukemia, Myeloid, Acute | interventions — Gemtuzumab

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: gemtuzumab ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; Mylotarg
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies gemtuzumab ozogamicin in treating patients with relapsed or refractory acute myeloid leukemia or acute promyelocytic leukemia. Monoclonal antibodies, such as gemtuzumab ozogamicin, can block cancer growth in different ways. Some block the ability of cancer to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To provide patients with acute myeloid leukemia (AML) or acute promyelocytic leukemia (APL), who have relapsed or who are refractory to standard treatments, with access to gemtuzumab ozogamicin (Mylotarg) when no other comparable or satisfactory alternative therapy is available.

II. To carefully monitor safety and to report safety information from patients receiving Mylotarg in this setting.

OUTLINE:

Patients receive gemtuzumab ozogamicin intravenously (IV) over 2 hours on days 1 and 15.

After completion of study treatment, patients are followed up every month for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed or refractory AML and not candidate for standard consolidation treatment after daunorubicin and cytosine arabinoside OR diagnosis of APL relapsed after tretinoin (ATRA) and arsenic trioxide therapy or APL with persisting or rising blasts, and no other comparable or satisfactory alternative therapy available (including patients not eligible for, or who have access to, investigational therapies via a clinical trial)
* Patients must have an initial diagnosis of AML, biphenotypic acute leukemia, or APL
* Patients must have cluster of differentiation (CD)33 positivity of > 30%
* Eastern Cooperative Oncology Group (ECOG) performance status =< 3 / Karnofsky > 60%
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2 x institutional upper limit of normal
* It is deemed ethical to provide an experimental drug (e.g., Mylotarg) that is associated with hepatotoxicity (veno-occlusive disease [VOD]) and myelosuppression
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to receiving Mylotarg and for the duration of treatment; should a woman become pregnant or suspect she is pregnant while receiving treatment with Mylotarg, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written Institutional Review Board (IRB)-approved informed consent document

Exclusion Criteria:

* Patients may not currently be receiving any other investigational agents for leukemia
* Patients with known untreated hepatitis C
* Uncontrolled intercurrent illness including, but not limited to active liver disease, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with Mylotarg
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients with a known hypersensitivity to gemtuzumab ozogamicin or its parts: recombinant humanized anti-CD33 monoclonal (hP67.6) antibody, calicheamicin derivatives or other ingredients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Ellis, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States